CLINICAL TRIAL: NCT02925156
Title: Modeling the Epidemiologic Transition: Energy Expenditure, Obesity and Diabetes
Brief Title: Modeling the Epidemiologic Transition Study
Acronym: METS
Status: Completed | Type: Observational
Sponsor: Loyola University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Amy Luke, Professor, Loyola University
Other Study IDs: 200038; R01DK080763 (NIH)
Record Dates: First submitted 2016-10-03; First posted 2016-10-05 (Estimated); Results first posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Obesity; Diabetes
Keywords: Activity Energy Expenditure; Doubly Labeled Water; Physical Activity; Obesity; Diabetes; Cardiovascular Disease; Adiponectin; Leptin; Ghrelin
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Motor Activity; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (10):
- Ghanaian Men: Men in the Ghana cohort are located at or near the the village of Nkwantakese which is approximately 20 kilometers outside of Kwame Nkrumah University of Science and Technology in Kumasi.
- South African Men: Men in the South Africa cohort are located at or near Khayelitsha, the 3rd largest township in South Africa, which is an adjacent town to the city of Cape Town. The population of Khayelitsha is about 500,000 people.
- Seychelles Men: Men in the Seychelles cohort are located at or near The Republic of Seychelles, which is an archipelago with 81,000 inhabitants located approximately 1,500 km east of Kenya in the Indian Ocean and approximately 2,000 km north of the island of Mauritius.
- Jamaican Men: Men in the Jamaica cohort are located at or near Spanish Town, Jamaica which is an urban area 25 km from the center of Kingston. The population of Spanish Town in 1991 was estimated at 92,000 people.
- United States Men: Men in the United States cohort are located at or near Maywood, IL, which is an African-American working class community adjacent to the western border of Chicago, IL. The population of Maywood in 2010 was estimated at 24,090 people.
- Ghanaian Women: Women in the Ghana cohort are located at or near the the village of Nkwantakese which is approximately 20 kilometers outside of Kwame Nkrumah University of Science and Technology in Kumasi.
- South African Women: Women in the South Africa cohort are located at or near Khayelitsha, the 3rd largest township in South Africa, which is an adjacent town to the city of Cape Town. The population of Khayelitsha is about 500,000 people.
- Seychelles Women: Women in the Seychelles cohort are located at or near The Republic of Seychelles, which is an archipelago with 81,000 inhabitants located approximately 1,500 km east of Kenya in the Indian Ocean and approximately 2,000 km north of the island of Mauritius.
- Jamaican Women: Women in the Jamaica cohort are located at or near Spanish Town, Jamaica which is an urban area 25 km from the center of Kingston. The population of Spanish Town in 1991 was estimated at 92,000 people.
- United States Women: Women in the United States cohort are located at or near Maywood, IL, which is an African-American working class community adjacent to the western border of Chicago, IL. The population of Maywood in 2010 was estimated at 24,090 people.

SUMMARY:
This project examines whether individuals' amount of activity energy expenditure (AEE) is related to adiposity and adiposity/diabetes-related hormones in a diverse sample of 2500, and to test the ecological hypothesis that a decline in levels of AEE is an important cause of the increases in obesity that are currently taking place in many societies.

One goal is to use doubly labeled water and/or accelerometers to objectively measure activity energy expenditure in community samples from five adult populations across the spectrum of obesity risk. From each site, (i.e., Ghana, South Africa, Seychelles, Jamaica, and the US), 500 black adults will be recruited. Among all participants, AEE will be measured using accelerometers and in a subset of 75 per site, AEE will also be measured by doubly labeled water.

The doubly labeled water sample will be used to confirm site-specific concordance with the accelerometer measurements and to estimate population mean levels of AEE. Additionally, body composition, dietary intake, fasting glucose, insulin, adiponectin, leptin and ghrelin will be measured. The relationships between calories expended in activity and body composition, dietary intake, glucose, hormones and adipocytokines, both within and between each population using doubly labeled water and accelerometers will be examined. In this longitudinal study, weight will be measured at 12 and 24-months, and AEE by accelerometer will be assessed at enrollment and again at 2-years of follow-up; associations between change in AEE and change in weight will be estimated.

The central purpose of this project is to test whether AEE or change in AEE can be identified as a contributory mechanism to population-wide weight gain and, if so, to quantify its importance. In addition, we seek to understand the interrelationships between the adipocytokines and the hormones ghrelin and insulin as well as AEE in the regulation of body weight across the continuum of body mass indices (BMI) represented by these five populations.

DETAILED DESCRIPTION:
Populations all over the world are experiencing rapid increases in the prevalence of obesity and diabetes. To date, the public health response to the emerging obesity epidemic has been almost totally ineffective. As a first line of response, professional bodies and government organizations have issued prevention guidelines, all of which include recommendations on levels of activity energy expenditure (AEE). However, even if fully implemented, it is not clear that the current recommendations on AEE would impact the trend in age-related weight gain. In fact, there is virtually no direct evidence that can be brought to bear on the question of whether the obesity epidemic has resulted primarily or even partially from society-wide declines in habitual physical activity (PA).

To date, epidemiologic research on AEE has relied on very crude measurement tools-primarily questionnaires. These self-reported data capture only a small fraction of the total variance in activity and are potentially confounded when they focus on leisure-time PA. By contrast, direct measurement with doubly labeled water (DLW) provides a precise, unbiased estimate of all forms of non-resting energy expenditure. DLW has also been used to validate the new generation of accelerometers which are efficient measurement tools for larger studies.

In this study, objective measurement tools will be used to examine the "ecology of AEE". This study will take place in 5 countries spanning the range of the activity-obesity spectrum and will combine both within-population person-level and between-population ecological analyses. First, the study will examine whether an individual's amount or pattern of AEE is related to adiposity in a diverse sample of 2,500. Second, the study will evaluate whether a decline in levels of AEE is an important cause of the rapid increases in obesity that currently take place in many societies. As an exploratory aim we will examine the role of selected adipocytokines and the appetite hormone ghrelin.

ELIGIBILITY:
Inclusion Criteria:

* Identify as African American or Black
* Age 18-50

Exclusion Criteria:

* Pregnancy, nursing, or planning to become pregnant
* Movement disorders or other disability that limits mobility

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study is comprises a complex samples population based approach drawn from communities in 5 countries: Ghana, Seychelles, South Africa, Jamaica and the US. Approximately 500 participants are enrolled per site for an unweighted total of 2500 participants.
Sampling Method: Non-Probability Sample
Enrollment: 2506 (Actual)
Dates: Start 2008-07-16 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Luke, PhD, Principal Investigator — Loyola University
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zimmet P. The burden of type 2 diabetes: are we doing enough? Diabetes Metab. 2003 Sep;29(4 Pt 2):6S9-18. doi: 10.1016/s1262-3636(03)72783-9. PMID 14502096
- [Background] Scaglione R, Argano C, Di Chiara T, Licata G. Obesity and cardiovascular risk: the new public health problem of worldwide proportions. Expert Rev Cardiovasc Ther. 2004 Mar;2(2):203-12. doi: 10.1586/14779072.2.2.203. PMID 15151469
- [Background] Popkin BM, Gordon-Larsen P. The nutrition transition: worldwide obesity dynamics and their determinants. Int J Obes Relat Metab Disord. 2004 Nov;28 Suppl 3:S2-9. doi: 10.1038/sj.ijo.0802804. PMID 15543214
- [Background] Kohn M, Booth M. The worldwide epidemic of obesity in adolescents. Adolesc Med. 2003 Feb;14(1):1-9. PMID 12529186
- [Background] James PT. Obesity: the worldwide epidemic. Clin Dermatol. 2004 Jul-Aug;22(4):276-80. doi: 10.1016/j.clindermatol.2004.01.010. PMID 15475226
- [Background] Pate RR, Pratt M, Blair SN, Haskell WL, Macera CA, Bouchard C, Buchner D, Ettinger W, Heath GW, King AC, et al. Physical activity and public health. A recommendation from the Centers for Disease Control and Prevention and the American College of Sports Medicine. JAMA. 1995 Feb 1;273(5):402-7. doi: 10.1001/jama.273.5.402. PMID 7823386
- [Background] Fletcher GF, Balady G, Blair SN, Blumenthal J, Caspersen C, Chaitman B, Epstein S, Sivarajan Froelicher ES, Froelicher VF, Pina IL, Pollock ML. Statement on exercise: benefits and recommendations for physical activity programs for all Americans. A statement for health professionals by the Committee on Exercise and Cardiac Rehabilitation of the Council on Clinical Cardiology, American Heart Association. Circulation. 1996 Aug 15;94(4):857-62. doi: 10.1161/01.cir.94.4.857. No abstract available. PMID 8772712
- [Background] Physical activity and cardiovascular health. NIH Consensus Development Panel on Physical Activity and Cardiovascular Health. JAMA. 1996 Jul 17;276(3):241-6. PMID 8667571
- [Background] Morrow JR Jr, Jackson AW, Bazzarre TL, Milne D, Blair SN. A one-year follow-up to physical activity and health. A report of the Surgeon General. Am J Prev Med. 1999 Jul;17(1):24-30. doi: 10.1016/s0749-3797(99)00030-6. PMID 10429749
- [Background] Trumbo P, Schlicker S, Yates AA, Poos M; Food and Nutrition Board of the Institute of Medicine, The National Academies. Dietary reference intakes for energy, carbohydrate, fiber, fat, fatty acids, cholesterol, protein and amino acids. J Am Diet Assoc. 2002 Nov;102(11):1621-30. doi: 10.1016/s0002-8223(02)90346-9. No abstract available. PMID 12449285
- [Result] Luke A, Bovet P, Plange-Rhule J, Forrester TE, Lambert EV, Schoeller DA, Dugas LR, Durazo-Arvizu RA, Shoham DA, Cao G, Brage S, Ekelund U, Cooper RS. A mixed ecologic-cohort comparison of physical activity & weight among young adults from five populations of African origin. BMC Public Health. 2014 Apr 24;14:397. doi: 10.1186/1471-2458-14-397. PMID 24758286
- [Result] Dugas LR, Kliethermes S, Plange-Rhule J, Tong L, Bovet P, Forrester TE, Lambert EV, Schoeller DA, Durazo-Arvizu RA, Shoham DA, Cao G, Brage S, Ekelund U, Cooper RS, Luke A. Accelerometer-measured physical activity is not associated with two-year weight change in African-origin adults from five diverse populations. PeerJ. 2017 Jan 19;5:e2902. doi: 10.7717/peerj.2902. eCollection 2017. PMID 28133575

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began on July 16, 2008 and ended on February 22, 2019
Period: Overall Study
Arm/Group | Ghanaian Men | South African Men | Jamaican Men | Seychelles Men | United States Men | Ghanaian Women | South African Women | Jamaican Women | Seychelles Women | United States Women
Started | 207 | 236 | 249 | 230 | 245 | 293 | 268 | 251 | 270 | 257
Completed | 180 | 183 | 198 | 171 | 156 | 186 | 234 | 215 | 197 | 223
Not Completed | 27 | 53 | 51 | 59 | 89 | 107 | 34 | 36 | 73 | 34
Not completed — Lost to Follow-up | 27 | 53 | 51 | 59 | 89 | 107 | 34 | 36 | 73 | 34

BASELINE CHARACTERISTICS:
Population: The baseline analysis population comprises all participants who signed an informed consent document
Groups:
- Total: Total of all reporting groups
Arm/Group | Ghanaian Men | South African Men | Jamaican Men | Seychelles Men | United States Men | Ghanaian Women | South African Women | Jamaican Women | Seychelles Women | United States Women | Total
Number analyzed (Participants) | 207 | 236 | 249 | 230 | 245 | 293 | 268 | 251 | 270 | 257 | 2506
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.6 (6.7) | 33.7 (5.6) | 34.0 (5.9) | 36.5 (5.1) | 35.6 (6.2) | 34.0 (6.6) | 33.1 (6.0) | 34.7 (6.2) | 35.8 (6.0) | 35.0 (6.3) | 34.7 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 293 | 268 | 251 | 270 | 257 | 1339
  Male | 207 | 236 | 249 | 230 | 245 | 0 | 0 | 0 | 0 | 0 | 1167
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 0 | 0 | 0 | 0 | 245 | 0 | 0 | 0 | 0 | 257 | 502
  Ghana | 207 | 0 | 0 | 0 | 0 | 293 | 0 | 0 | 0 | 0 | 500
  South Africa | 0 | 236 | 0 | 0 | 0 | 0 | 268 | 0 | 0 | 0 | 504
  Jamaica | 0 | 0 | 249 | 0 | 0 | 0 | 0 | 251 | 0 | 0 | 500
  Seychelles | 0 | 0 | 0 | 230 | 0 | 0 | 0 | 0 | 270 | 0 | 500
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 22.2 (2.7) | 22.4 (4.3) | 23.6 (4.5) | 26.5 (4.9) | 29.7 (7.5) | 25.5 (5.2) | 31.9 (8.2) | 29.5 (6.7) | 27.6 (6.2) | 34.1 (8.8) | 27.4 (7.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight
Description: The change in body weight (measured in kilograms) will be measured for participants 24 months after baseline.
Time Frame: 24 months
Population: The analysis population comprises participants who have a baseline and follow-up body weight recorded
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | Ghanaian Men | South African Men | Jamaican Men | Seychelles Men | United States Men | Ghanaian Women | South African Women | Jamaican Women | Seychelles Women | United States Women
Number analyzed (Participants) | 180 | 183 | 198 | 171 | 156 | 186 | 234 | 215 | 197 | 223
kilograms (kg) | 0.69 (3.15) | 0.76 (4.67) | 0.20 (3.90) | 0.81 (5.22) | 0.11 (5.99) | 1.94 (4.10) | 2.15 (6.82) | -0.11 (3.72) | 2.33 (4.27) | 0.08 (6.60)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 2 years
Arm/Group | Ghanaian Men | South African Men | Jamaican Men | Seychelles Men | United States Men | Ghanaian Women | South African Women | Jamaican Women | Seychelles Women | United States Women
All-Cause Mortality (participants affected / at risk) | 0/207 | 0/236 | 0/249 | 0/230 | 0/245 | 0/293 | 0/268 | 0/251 | 0/270 | 0/257
Serious Adverse Events (participants affected / at risk) | 0/207 | 0/236 | 0/249 | 0/230 | 0/245 | 0/293 | 0/268 | 0/251 | 0/270 | 0/257
Other Adverse Events (participants affected / at risk) | 0/207 | 0/236 | 0/249 | 0/230 | 0/245 | 0/293 | 0/268 | 0/251 | 0/270 | 0/257

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-05-27): https://cdn.clinicaltrials.gov/large-docs/56/NCT02925156/Prot_SAP_000.pdf
  • Informed Consent Form (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/56/NCT02925156/ICF_001.pdf